CLINICAL TRIAL: NCT01591681
Title: Reduction of Nocturnal Hypoglycemia by Using Predictive Algorithms and Pump Suspension: An Outpatient Pilot Feasibility and Efficacy Study
Brief Title: Outpatient Pump Shutoff Pilot Feasibility and Efficacy Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PSO3; 1R01DK085591-01 (NIH)
Record Dates: First submitted 2012-04-30; First posted 2012-05-04 (Estimated); Results first posted 2014-06-05 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Hypoglycemia; Continuous Glucose Monitoring; Pump Suspension
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pump suspension algorithm (Active Comparator): The study laptop will be running actively during the night and suspending the patient's pump if the algorithm predicts hypoglycemia based on the patient's continuous glucose sensor trend.
  Interventions: Device: Pump suspension
- Standard of Care (No Intervention): The control algorithm will run passively and not recommend control the patient's pump.

INTERVENTIONS:
Device: Pump suspension — The study laptop will communicate to the pump causing a suspension based on output from the algorithm which predicts hypoglycemia based on the continuous glucose sensor trend.
  Arms: Pump suspension algorithm

SUMMARY:
The purpose of this study is to see whether low blood sugar at night can be reduced by using a system that turns off the insulin pump automatically. The study system includes a combination continuous glucose monitor (CGM)/ insulin pump made by Medtronic MiniMed, Inc and a regular laptop computer that runs a computer program that predicts low blood sugar. It works by (1) measuring the glucose levels under the skin with a continuous glucose monitor, (2) using a computer program on a laptop to predict what will happen to the glucose level over the next 35-55 minutes, and (3) turning off the insulin pump when the computer program predicts that low blood sugar will occur.

This study has several phases and will take about 3 months for a patient to complete. Patients will use the Medtronic CGM with the Enlite sensor at home for 10-15 days to be sure that they are able and willing to use this system and to determine if they meet the investigators study criteria to proceed with the next phase of the study. Patients will be provided teaching on how to use CGM data in real time. If a patient is not using a Medtronic CGM already, the patient will first use one at home for 10-15 days to be sure that he/she is able and willing to use it. If a patient is already using a Medtronic CGM, then his/her most recent 10-15 days of data will be used to find out if he/she is eligible. Those who need to complete the CGM run-in phase will have an extra office visit for training.

If eligible to continue in the study, patients will need to use the study system for 5 nights at home so that the investigators can make sure they are able to use it correctly. After that, patients will be asked to use the study system each night for an additional 6 to 8 weeks. If the system is active and predicts that a patient's blood sugar will become low, the insulin pump will shut off for up to 2 hours.

The study will include about 45 individuals at 3 clinical centers in the United States and Canada.

DETAILED DESCRIPTION:
Patients who are eligible for the clinical trial initially will use a Medtronic Continuous Glucose Monitor (CGM) at home to verify that the subject is able to use the CGM and insert sensors. Subjects already using a Medtronic CGM will skip this phase, provided that the eligibility criteria for CGM use and the study are met.

Patients who meet criteria for sensor use and the study will then use the closed-loop system at home for 5 days to demonstrate their ability to use the system and submit study data to the Coordinating Center.

Patients who successfully demonstrate their ability to use the system at home as described above will be eligible for the randomized trial phase. This phase consists of use of the full system as an outpatient for approximately 42 nights:

* Each night the blood glucose level will be checked with the study home blood glucose (BG) meter and used to perform a calibration of the CGM. This calibration must occur no more than 90 minutes prior to activation of the system. NOTE: Patients will be instructed to calibrate the CGM per manufacturer guidelines.
* Then the system will be activated, linking the CGM and insulin pump to the computer at the bedside.
* A randomization schedule on the laptop will be used to determine whether the 'pump shut off' application will be active that night or not.
* Patients will be blinded as to whether the pump shut off is active when a session is initiated each night.
* There will not be an alarm if the pump shuts off. The CGM alarm will be set to 60 mg/dL (3.3 mmol/L). When a CGM alarm occurs, the patient will be asked to measure the blood glucose with a BG meter, if he/she is aware of the alarm.
* The time period for outcome assessment each night will be from the time the system is activated until it is turned off in the morning
* Pump shut off, when it occurs, will be for up to 2 hours. Multiple instances of pump suspension can occur if there are recurrent predictions of hypoglycemia during the night.
* Patients will be asked to check blood glucose with the study BG meter, blood ketones with the study ketone meter, and urine ketones with a ketone strip each morning prior to breakfast and enter the results on the study laptop. The patient will be instructed to contact the study physician if the blood glucose or ketone readings are out of an expected range. Patients will be contacted if these morning safety values are not reported as required or are out of range.
* Patients will be asked to record all overnight carbohydrate intake on the study laptop.
* Patients will be asked to perform periodic data uploads using the study laptop. Monitoring processes will ensure that the patient is contacted if these uploads do not occur as required, or if review of an upload reveals any extreme, prolonged episodes of low or high blood glucose readings, or elevated morning blood glucose, blood ketone, or urine ketone values.

Upon completion of the study, patients as well as study clinicians will be asked to complete a questionnaire regarding use of the study system.

There will be one follow-up visit after 21 days in the clinical trial and a second follow-up visit after the completion of 42 nights of successful study system use. A successful night of study system use is defined as use of the system for at least four hours. Phone contacts with the patients will be made once a week.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 1 diabetes and using daily insulin therapy for at least one year and an insulin infusion pump for at least 6 months
* Age >/= 15.0 - 45 years
* HbA1c </= 8.0%
* Availability of internet access for periodic upload of study data

Exclusion Criteria:

* Diabetic ketoacidosis in the past 3 months
* Hypoglycemic seizure or loss of consciousness in the past 6 months
* History of seizure disorder (except for hypoglycemic seizure)
* History of any heart disease including coronary artery disease, heart failure, or arrhythmiasCoronary artery disease or heart failure
* Cystic fibrosis
* Current use of oral/inhaled glucocorticoids, beta-blockers or other medications, which in the judgment of the investigator would be a contraindication to participation in the study.
* History of ongoing renal disease (other than microalbuminuria), or liver disease (Creatinine > 1.5 mg/dL (0.08 mmol/L))
* Medical or psychiatric condition that in the judgment of the investigator might interfere with the completion of the protocol such as:

  * Inpatient psychiatric treatment in the past 6 months
  * Uncontrolled adrenal disorder
  * Abuse of alcohol
* Pregnancy
* Liver disease as defined by an ALT greater than 3 times the upper limit of normal

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 49 (Actual)
Dates: Start 2012-11; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roy Beck, MD, Ph.D., Principal Investigator — Jaeb Center for Health Research; Bruce Buckingham, MD, Study Chair — Stanford University; John Lum, MS, Study Director — Jaeb Center for Health Research
Locations (3):
- United States (2):
  - Stanford University, Stanford, California
  - Barbara Davis Center for Childhood Diabetes, Aurora, Colorado
- St. Joseph's Health Care, London, Ontario, Canada

REFERENCES:
- [Result] Maahs DM, Calhoun P, Buckingham BA, Chase HP, Hramiak I, Lum J, Cameron F, Bequette BW, Aye T, Paul T, Slover R, Wadwa RP, Wilson DM, Kollman C, Beck RW; In Home Closed Loop Study Group. A randomized trial of a home system to reduce nocturnal hypoglycemia in type 1 diabetes. Diabetes Care. 2014 Jul;37(7):1885-91. doi: 10.2337/dc13-2159. Epub 2014 May 7. PMID 24804697
- [Derived] Wilson DM, Calhoun PM, Maahs DM, Chase HP, Messer L, Buckingham BA, Aye T, Clinton PK, Hramiak I, Kollman C, Beck RW; In Home Closed Loop Study Group. Factors associated with nocturnal hypoglycemia in at-risk adolescents and young adults with type 1 diabetes. Diabetes Technol Ther. 2015 Jun;17(6):385-91. doi: 10.1089/dia.2014.0342. Epub 2015 Mar 11. PMID 25761202

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at Stanford University (Stanford, CA), the Barbara Davis Center (Denver, CO), and St. Joseph's Health Care (London, ON). A total of 49 subjects were enrolled between November 1, 2012 and February 20, 2013. Forty-five participants age 15-45 years old with type 1 diabetes (median HbA1c 6.8%) completed the trial.
Pre-assignment Details: After the run-in phase, a 42-night randomized trial was conducted in which each night was randomly assigned to have either predictive low glucose suspend system active (intervention) or inactive (control) with half of the nights being intervention and half control nights.
Groups:
- Randomized Nights- Treatment or Control: Each study night will be randomized to have either Predictive Low Glucose Suspend or to be inactive (control). On nights randomized to the intervention treatment, the study laptop will be running actively during the night and suspending the patient's pump if the algorithm predicts hypoglycemia based on the patient's continuous glucose sensor trend. (Pump suspension : The study laptop will communicate to the pump causing suspension based on output from the algorithm which predicts hypoglycemia based on the continuous glucose sensor trend.) On control nights, the algorithm will run passively and not recommend suspensions or resumption to the patient's pump.
Period: Overall Study
Arm/Group | Randomized Nights- Treatment or Control
Started | 49
Completed | 45
Not Completed | 4
Not completed — Didn't meet min hypoglycemia requirement | 3
Not completed — Failed to use system during run-in | 1

BASELINE CHARACTERISTICS:
Population: There were 45 participants who could use the Continuous Glucose Monitoring device and met a minimum amount of nocturnal hypoglycemia as well as successfully completed the run-in phase of system use at home for 5 nights to verify the ability to use it properly.
Arm/Group | Randomized Nights- Treatment or Control
Number analyzed (Participants) | 45
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 30 [22 to 39]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 21
Race/Ethnicity, Customized [Number; unit: participants]
  White non-Hispanic | 42
  Hispanic | 2
  Black | 1
Weight [Median (Inter-Quartile Range); unit: kg] | 70 [62 to 85]
Height [Median (Inter-Quartile Range); unit: cm] | 172 [163 to 178]
Body-mass index [Median (Inter-Quartile Range); unit: kg/m^2] | 24 [22 to 27]
Glycated hemoglobin [Median (Inter-Quartile Range); unit: percent] | 6.8 [6.4 to 7.6]
Diabetes duration [Median (Inter-Quartile Range); unit: years] | 15 [12 to 26]
Daily insulin dose [Median (Inter-Quartile Range); unit: U/day] | 45 [32 to 60]
Daily insulin dose [Median (Inter-Quartile Range); unit: U/kg/day] | 0.64 [0.44 to 0.78]

OUTCOME MEASURES:

1. Primary Outcome: Hypoglycemia Outcome: Percentage of Nights With Sensor Glucose Value </=60 mg/dl
Description: Each night is categorized as to whether hypoglycemia occurred. Hypoglycemia is defined as the occurrence of one or more CGM glucose values ≤60 mg/dL. The percentage of hypoglycemic nights will be tabulated separately with versus without the closed-loop control system in use. A repeated measures logistic regression model will be used to compare intervention versus control nights accounting for correlated data from the same subject and adjusting for the baseline (bedtime) sensor glucose.
Time Frame: Overnight from system activation to deactivation in the morning upon awakening for 42 nights of system use
Measure: Number; unit: percentage of nights
Units Other Than Participants: Number of Nights Analyzed
Arm/Group | Pump Suspension Algorithm | Standard of Care
Number analyzed (Participants) | 45 | 45
Number analyzed (Number of Nights Analyzed) | 942 | 970
percentage of nights | 21 | 33
Statistical Analysis 1: Comparison: Pump Suspension Algorithm vs Standard of Care; Sample size was computed to be 45 participants using the system for 42 nights (21 nights with system active and 21 control nights) for a total of 1,890 nights in order to have 90% power with a type 1 error rate of 5% to reject the null hypothesis of no difference in nocturnal hypoglycemia assuming a true population rate of 30% of control nights and 15% of intervention nights with hypoglycemia after adjusting for the correlation from repeated nights and misclassification due to sensor inaccuracy; Test type: Superiority or Other; p < 0.001, Repeated measures regression model — The a priori threshold for statistical significance is 0.05; Repeated measures regression model was used accounting for correlated data from the same participant and for the overnight measures

2. Secondary Outcome: Percentage of Sensor Glucose Values 71 to 180 mg/dL
Description: The median percentages of the number of glucose values with values of 71-180 mg/dL overall.
Time Frame: Overnight from system activation to deactivation in the morning upon awakening for 42 nights of system use
Measure: Median (Inter-Quartile Range); unit: percentage glucose values
Units Other Than Participants: Number of Nights Analyzed
Arm/Group | Pump Suspension Algorithm | Standard of Care
Number analyzed (Participants) | 45 | 45
Number analyzed (Number of Nights Analyzed) | 942 | 970
percentage glucose values | 82 [54 to 99] | 75 [46 to 93]
Statistical Analysis 1: Comparison: Pump Suspension Algorithm vs Standard of Care; Test type: Superiority or Other; p < 0.001, repeated measures logistic regression — The a priori threshold for statistical significance is 0.05; Was used to test differences using mixed effects and a within subject autocorrelation structure to account for multiple nights from the same subject

3. Secondary Outcome: Percentage of Nights With a Sensor Glucose Value </= 70 mg/dL
Time Frame: Overnight from system activation to deactivation in the morning upon awakening for 42 nights of system use
Measure: Number; unit: percentage of nights
Units Other Than Participants: Number of Nights Analyzed
Arm/Group | Pump Suspension Algorithm | Standard of Care
Number analyzed (Participants) | 45 | 45
Number analyzed (Number of Nights Analyzed) | 942 | 970
percentage of nights | 32 | 45
Statistical Analysis 1: Comparison: Pump Suspension Algorithm vs Standard of Care; Test type: Superiority or Other; p < 0.001, Repeated measures regression model — The a priori threshold for statistical significance is 0.05; [statistical method as in outcome 1, analysis 1]

4. Secondary Outcome: Proportion of Nights With a Sensor Glucose Value </= 50 mg/dL
Time Frame: Overnight from system activation to deactivation in the morning upon awakening for 42 nights of system use
Measure: Number; unit: percentage of nights
Units Other Than Participants: Number of Nights Analyzed
Arm/Group | Pump Suspension Algorithm | Standard of Care
Number analyzed (Participants) | 45 | 45
Number analyzed (Number of Nights Analyzed) | 942 | 970
percentage of nights | 10 | 19
Statistical Analysis 1: Comparison: Pump Suspension Algorithm vs Standard of Care; Test type: Superiority or Other; p < 0.001, Repeated measures regression model — The a priori threshold for statistical significance is 0.05; [statistical method as in outcome 1, analysis 1]

5. Secondary Outcome: Median Morning Blood Glucose
Description: Measured with a study home blood glucose meter.
Time Frame: 42 mornings following night of system use
Measure: Median (Inter-Quartile Range); unit: mg/dl
Units Other Than Participants: Number of Mornings Analyzed
Arm/Group | Pump Suspension Algorithm | Standard of Care
Number analyzed (Participants) | 45 | 45
Number analyzed (Number of Mornings Analyzed) | 942 | 970
mg/dl | 144 [114 to 186] | 129 [96 to 173]
Statistical Analysis 1: Comparison: Pump Suspension Algorithm vs Standard of Care; Test type: Superiority or Other; p < 0.001, Repeated measures regression model — The a priori threshold for statistical significance is 0.05; [statistical method as in outcome 1, analysis 1]

6. Secondary Outcome: Percent of Mornings With Glucose >250 mg/dL
Description: Measured with a study home blood glucose meter.
Time Frame: 42 mornings following night of system use
Measure: Number; unit: percentage of mornings
Units Other Than Participants: Number of Mornings Analyzed
Arm/Group | Pump Suspension Algorithm | Standard of Care
Number analyzed (Participants) | 45 | 45
Number analyzed (Number of Mornings Analyzed) | 942 | 970
percentage of mornings | 6 | 6
Statistical Analysis 1: Comparison: Pump Suspension Algorithm vs Standard of Care; Test type: Superiority or Other; p = 0.71, repeated measures logistic regression — The a priori threshold for statistical significance is 0.05; [statistical method as in outcome 2, analysis 1]

7. Secondary Outcome: Percent of Mornings With Blood Ketones >1.0 mmol/L
Description: Blood ketones measured with a study blood ketone meter.
Time Frame: 42 mornings following night of system use
Measure: Number; unit: percentage of mornings
Units Other Than Participants: Number of Mornings Analyzed
Arm/Group | Pump Suspension Algorithm | Standard of Care
Number analyzed (Participants) | 45 | 45
Number analyzed (Number of Mornings Analyzed) | 942 | 970
percentage of mornings | 0.1 | 0.3
Statistical Analysis 1: Comparison: Pump Suspension Algorithm vs Standard of Care; Test type: Superiority or Other; p = 0.62, repeated measures logistic regression — The a priori threshold for statistical significance is 0.05; [statistical method as in outcome 2, analysis 1]

8. Secondary Outcome: Percent of Mornings With Urine Ketones >/= 15 mg/dl
Description: Urine ketones measured each morning with Ketostix.
Time Frame: 42 mornings following night of system use
Measure: Number; unit: percentage of mornings
Units Other Than Participants: Number of Mornings Analyzed
Arm/Group | Pump Suspension Algorithm | Standard of Care
Number analyzed (Participants) | 45 | 45
Number analyzed (Number of Mornings Analyzed) | 942 | 970
percentage of mornings | 3 | 2
Statistical Analysis 1: Comparison: Pump Suspension Algorithm vs Standard of Care; Test type: Superiority or Other; p = 0.10, repeated measures logistic regression — The a priori threshold for statistical significance is 0.05; [statistical method as in outcome 2, analysis 1]

9. Secondary Outcome: Overall Mean Sensor Glucose Overnight
Description: Calculated as the median of the overall mean.
Time Frame: Overnight from system activation to deactivation in the morning upon awakening for 42 nights of system use
Measure: Median (Inter-Quartile Range); unit: mg/dl
Units Other Than Participants: Number of Nights Analyzed
Arm/Group | Pump Suspension Algorithm | Standard of Care
Number analyzed (Participants) | 45 | 45
Number analyzed (Number of Nights Analyzed) | 942 | 970
mg/dl | 132 [110 to 163] | 125 [98 to 163]
Statistical Analysis 1: Comparison: Pump Suspension Algorithm vs Standard of Care; Test type: Superiority or Other; p < 0.001, Repeated measures regression model — The a priori threshold for statistical significance is 0.05; [statistical method as in outcome 1, analysis 1]

10. Secondary Outcome: Overnight Area Under the Curve 250 mg/dl Per 8 Hour
Description: The measure is reporting area under the curve for glucose concentrations below 250 mg/dL and above 60 mg/dL. Overall time below and above a threshold and area under a curve was divided by total time and multiplied by 8 hours.
Time Frame: Overnight from system activation to deactivation in the morning upon awakening for 42 nights of system use
Measure: Median (Inter-Quartile Range); unit: mg*hr/dL
Units Other Than Participants: Number of Nights Analyzed
Arm/Group | Pump Suspension Algorithm | Standard of Care
Number analyzed (Participants) | 45 | 45
Number analyzed (Number of Nights Analyzed) | 942 | 970
mg*hr/dL | 219 [72 to 666] | 236 [83 to 772]
Statistical Analysis 1: Comparison: Pump Suspension Algorithm vs Standard of Care; Test type: Superiority or Other; p = 0.98, Repeated measures regression model — The a priori threshold for statistical significance is 0.05; [statistical method as in outcome 1, analysis 1]

11. Secondary Outcome: Percent of Nights With Sensor Glucose >250 mg/dL
Time Frame: Overnight from system activation to deactivation in the morning upon awakening for 42 nights of system use
Measure: Number; unit: percentage of nights
Units Other Than Participants: Number of Nights Analyzed
Arm/Group | Pump Suspension Algorithm | Standard of Care
Number analyzed (Participants) | 45 | 45
Number analyzed (Number of Nights Analyzed) | 942 | 970
percentage of nights | 20 | 20
Statistical Analysis 1: Comparison: Pump Suspension Algorithm vs Standard of Care; Test type: Superiority or Other; p = 0.93, Repeated measures regression model — The a priori threshold for statistical significance is 0.05; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Groups:
- Pump Suspension Algorithm: Each study night will be randomized to have either Predictive Low Glucose Suspend or to be inactive (control). On nights randomized to the intervention treatment, the study laptop will be running actively during the night and suspending the patient's pump if the algorithm predicts hypoglycemia based on the patient's continuous glucose sensor trend. (Pump suspension : The study laptop will communicate to the pump causing suspension based on output from the algorithm which predicts hypoglycemia based on the continuous glucose sensor trend.)
- Standard of Care: On control nights, the algorithm will run passively and not recommend suspensions or resumption to the patient's pump.
Arm/Group | Pump Suspension Algorithm | Standard of Care
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 0/45 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No